CLINICAL TRIAL: NCT00139542
Title: Automated External Defibrillator (AED) Use in Out-of-Hospital Cardiac Arrest: A New Algorithm Named "One Shock Per Minute"
Brief Title: AED Use in Out-of-Hospital Cardiac Arrest: A New Algorithm Named "One Shock Per Minute"
Acronym: DEFI2005
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fire Brigade Of Paris Emergency Medicine Dept (Other)
Collaborators: Brigade de Sapeurs Pompiers de Paris (Unknown); Physio-Control, Inc, A division of Medtronic (Unknown)
Responsible Party: Daniel Jost, MD, Brigade de Sapeurs Pompiers de Paris
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BSPP01092005
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2009-05-11 (Estimated); Status verified 2009-05

CONDITIONS: Heart Arrest; Ventricular Fibrillation
Keywords: human; ventricular fibrillation; out-of-hospital; cardiac arrest; automated external defibrillators (AED); defibrillators; electrick countershock; cardiopulmonary resuscitation
MeSH Terms: conditions — Heart Arrest; Ventricular Fibrillation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CONTROL (Active Comparator): AED Treatment protocol following AHA Guidelines 2000 recommendations for cardiac arrest resuscitation.
  Interventions: Other: Guidelines 2000 AED protocol
- STUDY (Experimental): AED treatment protocol with prolonged CPR intervals, single shocks, fewer rhythm analysis and pulse checks.
  Interventions: Other: One shock per minute AED protocol

INTERVENTIONS:
Other: One shock per minute AED protocol — Single shocks; No post-shock pulse checks; 60 sec CPR before first shock; 30 sec CPR between rhythm analysis and shock delivery.
  Other Names: Biphasic LIFEPAK(R) 500 AED with cprMAX technology
  Arms: STUDY
Other: Guidelines 2000 AED protocol — Up to 3 consecutive shocks in a stack; No initial CPR prior to the first shock; Post-shock pulse checks after each non-shockable rhythm analysis; 60 sec CPR after each non-shockable rhythm analysis.
  Other Names: Biphasic LIFEPAK(R) 500 AED with cprMAX technology
  Arms: CONTROL

SUMMARY:
The aim of the trial is to evaluate a new AED algorithm that proposes a new timeline between the time devoted to administer a defibrillation shock, and the time devoted to chest compressions.

The researchers propose to decrease the periods of interruption of cardiopulmonary resuscitation (CPR), while keeping the principle of early defibrillation.

DETAILED DESCRIPTION:
Early use of semi-automated external defibrillators (AED) by Emergency Care teams in out-of-hospital cardiac arrest (OHCA), has been correlated with a significant gain in sequelae-free survival. The AED is programmed with an algorithm based recommended guidelines.

We will test a new algorithm that takes into account recent findings in pathophysiology.

Patients presenting with cardiovascular and pulmonary arrest treated by the BSPP Emergency Care who meet inclusion criterion are proposed for inclusion in the trial.

The aim of the trial is to evaluate a new AED algorithm that proposes a new timeline between the time devoted to administer a defibrillation shock, and the time devoted to chest compressions.

The new algorithm is entitled "one shock per minute". Use of this algorithm should validate several hypotheses:

* the importance of administering cardiac massage and artificial ventilation (CPR) prior to initiation of electrical shock treatment.
* the importance of continuing CPR immediately following electrical shock treatment
* the importance of reducing time between CPR procedures to a minimum
* the fact that three successive electrical shocks are of no therapeutic benefit.

We want to compare the control algorithm with the new one titled "one shock per minute", for shocked patients.

The sample size of this trial was calculated to provide a power of 85% and a type 1 error rate of alpha = 0.0294 for detecting an 11% increase in the rate of hospital admission, from its historical rate of 34% to a new rate of 45%. One interim analysis was planned with the stopping boundary alpha = 0.0294. This required inclusion of 430 patients in each group.

The primary endpoint is defined as "the admission of the patient alive at the hospital".

The secondary endpoints are defined as following :

- Detection of Palpable Carotid Pulse (ROSC) within the first 8 minutes after the connection of the AED The other secondary endpoint is survival to one year.

Concerning patients that do not receive shocks

They represent a priori 82% of the patients. The absolute number is a priori 3940, that is to say, 1970 in both two groups.

They will be used for an advanced observational descriptive study, to establish hypothesis for future studies.The same primary and secondary endpoints will be evaluated for them.

Among these patients not shocked, the algorithm foresees 60 seconds of CPR for the Control Group, and 90 seconds for the Trial Group. This setting relies on the hypothesis that increasing the time dedicated to chest compressions will increase the probability of return of a palpable pulse (ROSC), even for patients who do not fibrillate.

Statistical analysis will be completed by "Hôpital d'Instruction des Armées BEGIN - Epidemiology department"

We propose a comparison using the Chi square test for qualitative variables, Student's t test for quantitative variables, completion of a logistics model to analyze prognostic factors, as well as the proportional hazards model for survival analysis. Tests will be bilateral (significant p = 0,029 if we consider one intermediate analysis).

Overall analysis strategy will be defined and completed by the Epidemiology department of Hôpital d'Instruction des Armées BEGIN

ELIGIBILITY:
Inclusion Criteria:

* Patients in a state of apparent death as noted on arrival of the emergency care team vehicle
* Resuscitation by first aid team with a minimum of three people
* Analysis of cardiac rhythm by the AED possible
* At least one appropriate shock delivered by the AED

Exclusion Criteria:

* Many victims (>3) that must be treated simultaneously
* Signs of certain death (lividity)
* Patient with palpable pulse on arrival of emergency care team
* Patient already connected to another device
* Incident involving an AED that requires a "materiovigilance" report

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5107 (Actual)
Dates: Start 2005-09; Primary Completion 2007-03 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
the number of patients appropriately shocked by AED admitted alive at hospital / the total number of patients appropriately shocked by AED | within the first day after the first cardiac arrest

SECONDARY OUTCOMES:
Concerning patients appropriately shocked by AED: - return of spontaneous circulation (ROSC) at the arrival of physician on the scene | within the first hour after the first cardiac arrest
- ROSC within the first 8 minutes after the connection of the AED | within the 8 minutes after the connection of the AED
- Patient survival determined throughout the followup period of 1 year post-arrest. | one year after cardiac arrest
Safety endpoints were occurrences of CPR-related hemothorax requiring thoracic drain and/or hemorrhagic lesions requiring transfusion | within days of the cardiac arrest
Concerning patients not shocked by AED: - ROSC within the first 8 minutes after the connection of the AED | day of the cardiac arrest
- patient admitted alive to the hospital | within 24-48 hours of the cardiac arrest

CONTACTS AND LOCATIONS:
Overall Officials: Jost Daniel, Doctor, Principal Investigator — Fire Brigade of Paris
Locations (1):
- Fire Brigade of Paris Emergency medicine department, Paris, France

REFERENCES:
- [Background] Carpenter J, Rea TD, Murray JA, Kudenchuk PJ, Eisenberg MS. Defibrillation waveform and post-shock rhythm in out-of-hospital ventricular fibrillation cardiac arrest. Resuscitation. 2003 Nov;59(2):189-96. doi: 10.1016/s0300-9572(03)00183-7. PMID 14625109
- [Background] van Alem AP, Sanou BT, Koster RW. Interruption of cardiopulmonary resuscitation with the use of the automated external defibrillator in out-of-hospital cardiac arrest. Ann Emerg Med. 2003 Oct;42(4):449-57. doi: 10.1067/s0196-0644(03)00383-4. PMID 14520315
- [Background] Eisenberg MS, Horwood BT, Cummins RO, Reynolds-Haertle R, Hearne TR. Cardiac arrest and resuscitation: a tale of 29 cities. Ann Emerg Med. 1990 Feb;19(2):179-86. doi: 10.1016/s0196-0644(05)81805-0. PMID 2301797
- [Background] Cummins RO, Ornato JP, Thies WH, Pepe PE. Improving survival from sudden cardiac arrest: the "chain of survival" concept. A statement for health professionals from the Advanced Cardiac Life Support Subcommittee and the Emergency Cardiac Care Committee, American Heart Association. Circulation. 1991 May;83(5):1832-47. doi: 10.1161/01.cir.83.5.1832. No abstract available. PMID 2022039
- [Background] Jost D, Richter F, Morell E, Michel A, Goldstein P, Petit P et al. Expérience française de la défibrillation semi-automatique. Jeur, 1998;3:1A24-131.
- [Background] Cummins RO, Chamberlain DA, Abramson NS, Allen M, Baskett PJ, Becker L, Bossaert L, Delooz HH, Dick WF, Eisenberg MS, et al. Recommended guidelines for uniform reporting of data from out-of-hospital cardiac arrest: the Utstein Style. A statement for health professionals from a task force of the American Heart Association, the European Resuscitation Council, the Heart and Stroke Foundation of Canada, and the Australian Resuscitation Council. Circulation. 1991 Aug;84(2):960-75. doi: 10.1161/01.cir.84.2.960. No abstract available. PMID 1860248
- [Background] Halawa B. [Treatment of cardiac arrhythmia in pregnant women]. Pol Merkur Lekarski. 2000 Aug;9(50):513-8. Polish. PMID 11081313
- [Background] Sato Y, Weil MH, Sun S, Tang W, Xie J, Noc M, Bisera J. Adverse effects of interrupting precordial compression during cardiopulmonary resuscitation. Crit Care Med. 1997 May;25(5):733-6. doi: 10.1097/00003246-199705000-00005. PMID 9187589
- [Background] Cobb LA, Fahrenbruch CE, Walsh TR, Copass MK, Olsufka M, Breskin M, Hallstrom AP. Influence of cardiopulmonary resuscitation prior to defibrillation in patients with out-of-hospital ventricular fibrillation. JAMA. 1999 Apr 7;281(13):1182-8. doi: 10.1001/jama.281.13.1182. PMID 10199427
- [Background] Wik L, Hansen TB, Fylling F, Steen T, Vaagenes P, Auestad BH, Steen PA. Delaying defibrillation to give basic cardiopulmonary resuscitation to patients with out-of-hospital ventricular fibrillation: a randomized trial. JAMA. 2003 Mar 19;289(11):1389-95. doi: 10.1001/jama.289.11.1389. PMID 12636461
- [Background] Berg RA, Hilwig RW, Kern KB, Ewy GA. Precountershock cardiopulmonary resuscitation improves ventricular fibrillation median frequency and myocardial readiness for successful defibrillation from prolonged ventricular fibrillation: a randomized, controlled swine study. Ann Emerg Med. 2002 Dec;40(6):563-70. doi: 10.1067/mem.2002.129866. PMID 12447331
- [Background] Eftestol T, Sunde K, Steen PA. Effects of interrupting precordial compressions on the calculated probability of defibrillation success during out-of-hospital cardiac arrest. Circulation. 2002 May 14;105(19):2270-3. doi: 10.1161/01.cir.0000016362.42586.fe. PMID 12010909
- [Background] Banville I, Walker RG, Chapman FW. Maximizing CPR by changing the AED configuration. IICE2005 Book of Abstracts; p 26.
- [Background] Jost D, Calamai F, Fontaine D et al. Concordance Between Carotid Pulse Check and Transthoracic Impedance Characteristics in Out-of-Hospital Cardiac Arrest [abstr]. Circulation 2006;114:II_1201-a.
- [Background] Renard A, Jost D, Verret C et al. Effect of Thrombolytics on the Immediate Prognosis for Out-of-Hospital Cardiac Arrest [abstr]. Circulation 2007;116:II_928-b.
- [Result] Hersan O, Jost D, Banville IL et al. More CPR With the New Guidelines. Does It Impact VF Termination by Defibrillation Shocks? [abstr]. Circulation 2007;116:II_386-a.
- [Result] Jost D, Degrange H, Hersan O, Briche F, Fontaine D, Lallement D, Calamai F, Verret C, Banville I, Chapman F, Koster R, Descatha A, Petit J-L, Fuilla C. Prospective Clinical Trial, DEFI 2005: Does an AED Algorithm with More CPR Impact Out-of-Hospital Cardiac Arrest Prognosis? Resuscitation 2008;77 (Supp 1):.S18. (Abstract). ERC 2008
- [Result] Jost D, Banville I, Degrange H, Hersan O, Briche F, Dubourdieu S, Fontaine D, Lallement D, Chapman F, Lank P, Petit J-L, Fuilla C. Metronome Use to Improve CPR by Firefighters during Out-of-Hospital Cardiac Arrest. Academic Emergency Medicine 2008;15(s1):S21-S22. (Abstract). SAEM 2008.
- [Result] Jost D, Degrange H, Hersan O, Briche F, Fontaine D, Lallement D, Calamai F, Verret C, Banville I, Chapman F, Koster R, Fuilla C, Jost D, Descatha A, Dubourdieu S, Petit J-L, Lank P. Prospective Clinical Trial, DEFI 2005: Does an AED Algorithm with More CPR Impact Out-of-Hospital Cardiac Arrest Prognosis? Academic Emergency Medicine 2008;15(s1):S224-S225. (Abstract). SAEM 2008.
- [Result] Jost D, Banville I, Girardeau S, Calamai F, Fontaine D, Lallement D, Chapman FW, Degrange H, Petit J-L, Fuilla C. Impact of reducing CPR hands-off time during out-of-hospital cardiac arrest on post-shock rhythm progression. Eur Heart J. 2008;29:642 (Abstract).
- [Result] Jost D, Degrange H, Banville IL, Hersan O, Briche F, Fontaine D, Lallement D, Calamai F, Chapman FW, Petit J-L, Fuilla C. Is the Outcome from Witnessed VF Cardiac Arrest Improved by Providing More CPR? Results from DEFI2005, a Randomized Controlled Trial of two AED Protocols. Circulation. 2008;118:S_1447. (Abstract). AHA 2008
- [Derived] Jost D, Degrange H, Verret C, Hersan O, Banville IL, Chapman FW, Lank P, Petit JL, Fuilla C, Migliani R, Carpentier JP; DEFI 2005 Work Group. DEFI 2005: a randomized controlled trial of the effect of automated external defibrillator cardiopulmonary resuscitation protocol on outcome from out-of-hospital cardiac arrest. Circulation. 2010 Apr 13;121(14):1614-22. doi: 10.1161/CIRCULATIONAHA.109.878389. Epub 2010 Mar 29. PMID 20351239
- See also: This is the official Paris Fire Brigade website — http://www.pompiersparis.fr